CLINICAL TRIAL: NCT05881135
Title: Supplemental Citicoline Administration to Reduce Lung Injury Efficacy Trial (SCARLET)
Acronym: SCARLET
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Elliott Crouser, Professor of Internal Medicine, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022H0451
Record Dates: First submitted 2023-04-25; First posted 2023-05-31 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Cytidine Diphosphate Choline; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- IV 1 mg/kg/day Citicoline (Experimental): i.v. bolus of 10 ml normal saline containing citicoline 1 mg/kg, administered twice daily for 5 days.
  Interventions: Drug: Citicoline
- IV 5 mg/kg/day Citicoline (Experimental): i.v. bolus of 10 ml normal saline containing 5 mg/kg citicoline, administered twice daily for 5 days.
  Interventions: Drug: Citicoline
- IV 10 mg/kg/day Citicoline (Experimental): i.v. bolus of 10 ml normal saline containing 10 mg/kg citicoline, administered twice daily for 5 days.
  Interventions: Drug: Citicoline
- IV 10 ml normal saline (Placebo Comparator): i.v. bolus of 10 ml normal saline (without active ingredient) administered i.v., twice daily for 5 days.
  Interventions: Drug: Saline/Placebo

INTERVENTIONS:
Drug: Citicoline — i.v. bolus administration every 12 hours for 5 days.
  Other Names: Somazina, CDP-choline
  Arms: IV 1 mg/kg/day Citicoline; IV 10 mg/kg/day Citicoline; IV 5 mg/kg/day Citicoline
Drug: Saline/Placebo — i.v. administered every 12 hours as a 10 ml bolus for 5 days.
  Other Names: Normal saline solution
  Arms: IV 10 ml normal saline

SUMMARY:
The goal of this single center, double-blinded, placebo-controlled, and randomized Phase 1 trial is to determine if i.v. citicoline is safe and efficacious compared to i.v. saline/control in adults presenting with SARS CoV-2 infection complicated by acute hypoxemic respiratory failure. The main questions it aims to answer:

* Is citicoline safe in this patient population?
* Does citicoline have a benefit in terms of improving oxygenation?
* Does citicoline reduce overall severity of illness as reflected by standardized scales.

Patients will be assigned to i.v. treatment with citicoline or saline twice daily for 5 consecutive days. SpO2/FiO2 ratios will be recorded daily as per standard clinical practice to compare citicoline treatments at three different doses to placebo.

DETAILED DESCRIPTION:
SCARLET is a single center, double-blinded, placebo-controlled, and randomized Phase 1 trial of i.v. citicoline in adult patients of any sex, gender, age, or ethnicity who are present with acute hypoxemic respiratory failure due to SARS CoV-2 infection. The goals are safety over a range of doses based on the number of treatment related adverse events as assessed by CTCAE v.5, and demonstration of efficacy as reflected by SpO2/FiO2 measured at day 3 in hospitalized COVID infected patients with acute hypoxemic respiratory failure, as defined by requiring at least 4 liters nasal cannula oxygen supplementation to maintain the SpO2 above 90%. The trial will enroll 20 patients per dose for 3 citicoline doses (1, 5, and 10 mg/kg/day) along with 20 placebo-treated controls.

ELIGIBILITY:
1. The subject or their authorized representative must be able to understand and provide informed consent
2. Adult patients (≥18 years)
3. Laboratory-confirmed SARS-CoV-2 infection within the 10 days prior to randomization
4. Admitted to OSU East or OSU Main for acute respiratory failure (on at least 4 LPM oxygen)
5. C-reactive protein (CRP) > 32 mg/l
6. Adequate i.v. access available (either peripheral or central venous access)
7. Female subjects of childbearing potential must have a negative pregnancy test upon study entry

Exclusion Criteria:

1. Subjects who are unable or unwilling to give written informed consent or to comply with study protocol and who have no legal authorized representative available to give consent on their behalf
2. Individuals being treated with extracorporeal membrane oxygenation (ECMO)
3. Subjects who, in the clinicians estimation, will be unlikely to survive the protocol duration due to imminent and unavoidable risk of death
4. Individuals with hypertonia of the parasympathetic nervous system
5. Prisoners
6. Children (<18 years)
7. Women who may be pregnant, are pregnant, or have plans to become pregnant
8. Women who are breast feeding
9. Individuals with a known allergy to citicoline
10. Subjects that are taking medications that contain L-Dopa, centrophenoxine, or meclofenoxate
11. Subjects with past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the principal investigator (PI), may pose additional risks from participation in the study or that may impact the quality or interpretation of the data obtained from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-06-06 (Actual); Primary Completion 2025-03-17 (Actual); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Safety of citicoline over a range of doses in COVID-19 patients presenting with acute hypoxemic respiratory failure. | Until hospital discharge or up to 29 days
  Safety will be assessed in each arm of the study: 1, 5, or 10 mg/kg/day citicoline by i.v. bolus or i.v. saline bolus for 5 consecutive days. Safety analysis will be performed based on a continuous safety monitoring rule to guide accrual suspension decisions based on number of treatment-related adverse events as assessed by the CTCAE v.5.0. The number of patients with an SAE that would warrant temporary suspension of accrual in a given group corresponds to a high posterior probability that the true SAE probability is greater than an acceptable level (i.e., Pr(pi > 0.25 | data) > 0.85), where the posterior probability is determined from a Beta-Binomial distribution with Beta (1, 1) as the prior on pi.
Citicoline's effect on acute hypoxemic respiratory failure in COVID-19 patients. | Day 3
  The primary clinical outcome will be measured on Day 3: lowest recorded SpO2/FiO2 ratio.

SECONDARY OUTCOMES:
Effect of citicoline on COVID specific disease severity scale in patients with acute COVID associated hypoxemic respiratory failure. | Through day 8
  Days 1,3,5 and 8 COVID ordinal outcomes scale (COOS). The COOS scale ranges from 0-8 with higher scores corresponding with worse clinical outcomes.
Effect of citicoline on Sequential Organ Failure Score (SOFA) in patients with COVID associated acute respiratory failure. | Through day 8
  Days 1,3,5, and 8 composite and component SOFA scores measure while the study subject is in the ICU. SOFA scores range from 0-24 with higher scores corresponding to more severe organ failures.

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pannu S, Exline MC, Bednash JS, Englert JA, Diaz P, Bartlett A, Brock G, Wu Q, Davis IC, Crouser ED. SCARLET (Supplemental Citicoline Administration to Reduce Lung injury Efficacy Trial): study protocol for a single-site, double-blinded, placebo-controlled, and randomized Phase 1/2 trial of i.v. citicoline (CDP-choline) in hospitalized SARS CoV-2-infected patients with hypoxemic acute respiratory failure. Trials. 2024 May 18;25(1):328. doi: 10.1186/s13063-024-08155-0. PMID 38760804